CLINICAL TRIAL: NCT03818152
Title: Reliability and Validity of Strength Measurements of the Lower Limbs in Children With Bilateral Spastic Cerebral Palsy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B670201834766/Amendement
Record Dates: First submitted 2019-01-25; First posted 2019-01-28 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Children; Cerebral Palsy; Muscle Weakness
Keywords: Cerebral palsy; Children; Functional strength measurement; Lower limbs; Reproducability
MeSH Terms: conditions — Cerebral Palsy; Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Other): Reliability study isokinetic strength assessment of the lower limbs.
  Interventions: Other: Functional strength assessment

INTERVENTIONS:
Other: Functional strength assessment — Functional strength exercises to assess strength in lower limbs.

SUMMARY:
Specific musculo-tendinous adaptations in children with cerebral palsy (CP) have an influence on muscle strength and consequently on functional behavior and participation. Evidence of strength training programs has been shown on level of body function but transfer to levels of activity and participation is still limited. Lack of transfer is related to lack of specificity of the training and poor overall quality of the interventions (intensity, duration, frequency and/or type).

The use of functional strength exercises to assess and train strength of the lower limbs in children with CP is well implemented in the most functional children with CP (GMFCS-level I). To assess isometric strength the hand held dynamometer (HHD) can be used in clinical settings but reliability of this tool is questionable.

The aim of this study is to adapt existing functional strength tests for less functional children with CP (focussing on GMFCS level II and III) and to investigate the correlation with isometric strength measurements and other functional parameters.

DETAILED DESCRIPTION:
Specific musculo-tendinous adaptations in children with cerebral palsy (CP) have an influence on muscle strength and consequently on functional behavior and participation. Evidence of strength training programs has been shown on level of body function but transfer to levels of activity and participation is still limited. Lack of transfer is related to lack of specificity of the training and poor overall quality of the interventions (intensity, duration, frequency and/or type).

The use of functional strength exercises to assess and train strength of the lower limbs in children with CP is well implemented in the most functional children with CP (GMFCS-level I).

The aim of this study is to adapt existing functional strength tests for less functional children with CP (focussing on GMFCS-level II and III) and to investigate the correlation with isometric strength measurements and other functional parameters.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral spastic CP
* GMFCS II-III
* 6-18 Y
* No botox until 4 months before testing
* No orthopedic surgery until 1 Y before testing
* Good cooperation

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Functional testing | 60 minutes
  30 seconds tests (nr/30 seconds): the children have to perform as much as trials as possible within 30 seconds; e.g. stand up and sit

SECONDARY OUTCOMES:
Isometric strength test | 60 minutes
  Strength of the lower limbs (Nm) by means of a fixed hand held dynamometer
Core stability test | 30 minutes
  30 seconds tests (nr/3 30 seconds test (nr/30 seconds)
Gait capacity | 1 minute
  1 Minute Walking Test (m/1 minute)
Gait capacity | 5 minutes
  Timed up and go (seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided